CLINICAL TRIAL: NCT00143026
Title: Study to Compare the Effect of Treatment With Carbidopa/Levodopa/Entacapone on the Quality of Life of Patients With Parkinson's Disease.
Brief Title: Study to Compare the Effect of Treatment With Carbidopa/Levodopa/Entacapone on the Quality of Life of Patients With Parkinson's Disease. This Study is Not Recruiting in the United States
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CELC200A2406
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, levodopa, motor fluctuations
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo

INTERVENTIONS:
Drug: carbidopa, levodopa, entacapone

SUMMARY:
This study examines the effect of treatment of levodopa/entacapone on quality of life, as measured by the Parkinson's Disease-Questionnaire 8 (PDQ-8), in Parkinson's disease patients with no or minimal, non-disabling motor fluctuations.

DETAILED DESCRIPTION:
This study examines the effect of treatment of levodopa/entacapone on quality of life, as measured by the Parkinson's Disease-Questionnaire 8 (PDQ-8), in Parkinson's disease patients with no or minimal, non-disabling motor fluctuations. Treatment with carbidopa/levodopa/entacapone will be compared with treatment with standard formulation levodopa/carbidopa.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease exhibiting at least 2 or 3 symptoms
* Motor functions must be regarded as non-disabling by the patient

Exclusion Criteria:

* History, signs or symptoms suggesting the diagnosis of atypical or secondary parkinsonism
* History of dyskinesia
* Previous or current use of entacapone or tolcapone
* Unstable Parkinson's disease patients requiring/receiving regimens of levodopa
* Subjects taking levodopa/DDCI controlled release or extended release formulations

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment

SECONDARY OUTCOMES:
Symptom control change from baseline
Change from baseline in number of wearing-off symptoms
Change from baseline in proportion of patients experiencing wearing-off

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair
Locations (18):
- Australia (9):
  - Royal Adelaide Hospital, Adelaide
  - Watkins Medical Center, Brisbane
  - Central Coast Neuroscience Research, Gosford
  - Heidelberg Repatriation Hospital, Melbourne
  - Monash Medical Centre, Melbourne
  - Sir Charles Gairdner Hospital, Perth
  - Concord Hospital, Sydney
  - Southern Neurology, St. George Private Hospital, Sydney
  - Westmead Hospital, Sydney
- Philippines (2):
  - St. Luke's Medical Centre, Manila
  - University of Santo Tomas Hospital, Manila
- Taiwan (3):
  - Chang Gung Memorial Hospital, Linkou District
  - Kaohsiung Medical University, Chung-Ho Memorial Hospital, Linkou District
  - National Taiwan University Hospital, Linkou District
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Bangkok
  - Pharmongkutklao Army Hospital, Bangkok
  - Siriraj Hospital, Bangkok